CLINICAL TRIAL: NCT04281485
Title: A PHASE 3, MULTICENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO CONTROLLED STUDY TO EVALUATE THE SAFETY AND EFFICACY OF PF 06939926 FOR THE TREATMENT OF DUCHENNE MUSCULAR DYSTROPHY
Brief Title: Study to Evaluate the Safety and Efficacy of PF-06939926 for the Treatment of Duchenne Muscular Dystrophy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3391003; 2023-508510-42-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2020-02-11; First posted 2020-02-24 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Clinical trial; Gene therapy; Duchenne muscular dystrophy; fordadistrogene movaparvovec
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: Parallel up to the measurement of the primary outcome at Week 52. At the beginning of study Year 2 participants who were originally assigned to placebo will have the opportunity to receive PF-06939926. All participants will be followed for 5 years following treatment with PF-06939926.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be quadruple blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Other): Approximately two thirds of participants will be randomized to Cohort 1.
  Interventions: Genetic: PF-06939926; Other: Placebo
- Cohort 2 (Other): Approximately one third of participants will be randomized to Cohort 2.
  Interventions: Other: Placebo; Genetic: PF-06939926

INTERVENTIONS:
Genetic: PF-06939926 — PF-06939926 will be administered as a single IV infusion at Year 1 for Cohort 1.
  Arms: Cohort 1
Other: Placebo — Placebo will be administered as a single IV infusion at Year 1 for Cohort 2.
  Arms: Cohort 2
Other: Placebo — Placebo will be administered as a single IV infusion at Year 2 for Cohort 1.
  Arms: Cohort 1
Genetic: PF-06939926 — PF-06939926 will be administered as a single IV infusion at Year 2 for Cohort 2
  Arms: Cohort 2

SUMMARY:
The study will evaluate the safety and efficacy of gene therapy in boys with DMD. It is a randomized, double-blind, placebo-controlled study with two thirds of participants assigned to gene therapy. The one third of participants who are randomized to the placebo arm will have an opportunity for treatment with gene therapy at the beginning of the second year.

DETAILED DESCRIPTION:
The study will assess the efficacy of PF-06939926 gene therapy on ambulatory function while also monitoring its safety. Approximately 99 boys with DMD will be enrolled and randomly assigned to one of two groups: approximately two thirds will be in Cohort 1 and receive gene therapy at the start of the study; approximately one third will be in Cohort 2 and receive placebo at the start of the study and receive gene therapy after one year, as long as it remains safe to do so. The treatment (PF-06939926 gene therapy or placebo) will be given as an intravenous infusion lasting up to 2 hours.

The study includes boys who are at least 4 years old and less than 8 years old (including 7 year olds up until their 8th birthday). All boys will need to be on a daily dose of glucocorticoids (prednisone, prednisolone, or deflazacort) for at least 3 months prior to enrolling and to stay on daily glucocorticoids for the first 2 years of the study. All boys will need to be negative for neutralizing antibodies against AAV9, as measured by the test done for the study as part of screening.

The primary outcome of the study will be assessed at 52 weeks. All participants will be followed in the study for 15 years after treatment with gene therapy. Participants who received fordadistrogene movaparvovec in Pfizer studies C3391001 and C3391008 or are currently enrolled in Pfizer study C3391011 will be allowed to roll over into the long-term safety follow-up period of this study and will be considered Cohort 3.

The study medication, all medical tests associated with the study, and the visits to the study sites are free of charge. Participants will also be supported for travel costs associated with study visits.

ELIGIBILITY:
Key inclusion criteria:

1. Confirmed diagnosis of Duchenne muscular dystrophy by prior genetic testing
2. Receiving a stable daily dose (at least 0.5 mg/kg/day prednisone or prednisolone, or at least 0.75 mg/kg/day deflazacort) for at least 3 months prior to Screening
3. Ambulatory, as assessed by protocol-specified criteria

Key exclusion criteria:

1. Positive test performed by Pfizer for neutralizing antibodies to AAV9
2. Any treatment designed to increase dystrophin expression within 6 months prior to screening (e.g., Translarna™, EXONDYS 51™, VYONDYS 53™)
3. Any prior treatment with gene therapy
4. Any non-healed injury that may impact functional testing (eg NSAA)
5. Abnormality in specified laboratory tests, including blood counts, liver and kidney function
6. Any of the following genetic abnormalities in the dystrophin gene:

   1. Any mutation (exon deletion, exon duplication, insertion, or point mutation) affecting any exon between exon 9 and exon 13, inclusive; OR
   2. A deletion that affects both exon 29 and exon 30;OR
   3. A deletion that affects any exons between 56-71, inclusive.

Ages: 4 Years to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male
Enrollment: 114 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2039-04-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- United States (17):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Arkansas Children's, Little Rock, Arkansas
  - UCLA Medical Center, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - KU Clinical Research Center - Clinical and Translational Science Unit (CTSU) - Fairway, Fairway, Kansas
  - KU Clinical Research Center - Clinical and Translational Science Unit (CTSU) - Rainbow, Kansas City, Kansas
  - University of Kansas Hospital - Investigational Pharmacy, Kansas City, Kansas
  - University of Kansas Hospital - Pediatric and Pediatric ICU - Operating Room, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Pediatric Cardiology, Prairie Village, Kansas
  - Lenox Baker Children's Hospital, Durham, North Carolina
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Primary Childrens Hospital, Salt Lake City, Utah
  - University of Utah Clinical Neurosciences Center, Salt Lake City, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - Seattle Children's, Seattle, Washington
- Australia (3):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - The Royal Children's Hospital Melbourne, Parkville, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia
- Belgium (2):
  - UZ Gent, Ghent
  - UZ leuven, Leuven
- Canada (4):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's Hospital - London Health Sciences Centre, London, Ontario
  - Childrens Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital For Sick Children, Toronto, Ontario
- France (2):
  - CHU de Nantes- Hotel Dieu, Nantes
  - Hopital Necker, Paris
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitatsklinikum Essen, Essen
- Israel (2):
  - Hadassah University Medical Center, Ein Kerem, Jerusalem
  - Schneider Children's Medical Center of Israel, Petach Tikvah
- Italy (2):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - IRCCS Ospedale Pediatrico Bambino Gesù, Rome
- Japan (3):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Hyogo College of Medicine College Hospital, Nishinomiya, Hyōgo
  - National Center of Neurology and Psychiatry, Tokyo
- Russia (2):
  - Saint Petersburg State Paediatric Medical University, Saint Petersburg
  - State Autonomous Healthcare Institution of Sverdlovsk Region Children's City Clinical Hospital No 9, Yekaterinburg
- South Korea (3):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Switzerland (2):
  - Inselspital, University Children's Hospital Berne, Bern
  - Universitaets-Kinderspital Zuerich, Zurich
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (3):
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Alder Hey Children's NHS Foundation Trust, Liverpool, Merseyside
  - Great Ormond Street Institute of Child Health, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3391003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 114 participants were enrolled and received at least one dose of study treatment. Results are reported based on primary completion date of Week 52.
Pre-assignment Details: Primary Completion Date (PCD) defined as the time point when at least 90 randomized participants received investigational product and completed the one-year follow-up/week 52 visit.
Groups:
- Cohort 1: Participants were randomized to receive a single dose of fordadistrogene Movaparvovec 2*10^14 (2E14) vector genomes per kilogram body weight (vg/kg) on Day 1 (Year 1 Day 1) and a single dose of matching placebo on Day 390 (Year 2 Day 1).
- Cohort 2: Participants were randomized to receive a single dose of matching placebo on Day 1 (Year 1 Day 1) and a single dose of fordadistrogene Movaparvovec 2E14 vg/kg on Day 390 (Year 2 Day 1).
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 79 | 35
Received Treatment Year 1 Day 1 | 79 | 35
Received Treatment Year 2 Day 1 | 42 | 18
Completed (Completed indicates participants completed the Week 52 as of PCD) | 69 | 28
Not Completed | 10 | 7
Not completed — No Longer Met Eligibility Criteria | 0 | 2
Not completed — Ongoing (Safety data collection) | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Participants were randomized to receive a single dose of fordadistrogene Movaparvovec 2E14 vg/kg on Day 1 (Year 1 Day 1) and a single dose of matching placebo on Day 390 (Year 2 Day 1).
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 79 | 35 | 114
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.4 (1.3) | 6.6 (1.2) | 6.4 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 79 | 35 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 4 | 19
  Not Hispanic or Latino | 63 | 30 | 93
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 24 | 9 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 49 | 24 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in North Star Ambulatory Assessment (NSAA) Total Score at Week 52
Description: The NSAA was a 17-item test that graded performance of various functional skills using the following scale: 0 (unable to achieve independently), 1 (modified method but achieves goal independent of physical assistance from another), and 2 ("normal"- no obvious modification of activity). Total score was calculated as the sum of all 17 individual item responses and ranged from 0 (worst) to 34 (fully independent function) with higher scores indicating better function. Baseline NSAA total score is defined as the last non-missing NSAA total score collected prior to Year 1 drug administration.
Time Frame: Baseline, Week 52
Population: Full analysis set (FAS) through Week 52 included all eligible participants who were randomly assigned and received a single dose of study drug on Day 1 (Year 1 Day 1). Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 63 | 26
Score on a scale | 1.46 [0.61 to 2.30] | 1.37 [0.08 to 2.67]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2; Test type: Superiority; p = 0.9116, Mixed Models Analysis; Least Square Mean Difference = 0.09, 95% CI 2-sided [-1.46 to 1.64], Standard Error of Mean 0.78; The Mixed Model Repeated Measures (MMRM) model contained fixed effects for treatment group (categorical variable), visit (ordered categorical variable), and treatment group by visit interaction with additional fixed effects for baseline value (continuous variable), screening age (continuous variable), baseline value by visit interaction, and screening age by visit interaction with an unstructured variance-covariance matrix

2. Secondary Outcome: Change From Baseline in Percent Normal Dystrophin Expression Level in Muscle Biopsies by Liquid Chromatography Mass Spectrometry (LC-MS) Based on LLQV Peptide at Week 52
Description: The LC-MS assay measured the LLQVAVEDR (LLQV) peptide that detected full-length endogenous dystrophin as well as the mini-dystrophin transgene protein.
Time Frame: Baseline, Week 52
Population: FAS through Week 52 included all eligible participants who were randomly assigned and received a single dose of study drug on Day 1 (Year 1 Day 1). Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: % normal dystrophin expression level
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 11 | 7
% normal dystrophin expression level | 85.88 [63.09 to 108.67] | 0.13 [-28.46 to 28.72]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2; Test type: Superiority; p = 0.0002, ANCOVA; The ANCOVA model contained treatment group (categorical variable) and screening age (continuous variable); Least Square Mean Difference = 85.75, 95% CI 2-sided [49.15 to 122.35], Standard Error of Mean 17.17

3. Secondary Outcome: Change From Baseline in Percent of Muscle Fibers Expressing Mini-Dystrophin in Muscle Biopsies by Immunofluorescence at Week 52
Description: Muscle fibers expressing mini-dystrophin transgene protein were evaluated by immunofluorescent staining using the mini-dystrophin specific antibody which only recognized the mini-dystrophin transgene protein.
Time Frame: Baseline, Week 52
Population: FAS included all eligible participants who were randomly assigned and received a single dose of study drug on Day 1 (Year 1 Day 1). Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of muscle fibers
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 12 | 8
Percentage of muscle fibers | 50.15 [37.48 to 62.81] | -1.31 [-16.82 to 14.20]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2; Test type: Superiority; p < 0.0001, ANCOVA; The ANCOVA model contained treatment group (categorical variable) and screening age (continuous variable); Least Square Mean Difference = 51.46, 95% CI 2-sided [31.43 to 71.49], Standard Error of Mean 9.49

4. Secondary Outcome: Change From Baseline in Serum Creatine Kinase (CK) Concentration at Week 52
Description: The CK results were analyzed by the central laboratory.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Units per Liter (U/L)
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 60 | 23
Units per Liter (U/L) | 0.68 [0.60 to 0.77] | 1.06 [0.87 to 1.29]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Geometric Ratio of LS Means = 0.64, 95% CI 2-sided [0.50 to 0.81]; MMRM approach for log transformed data including visits through Week 52 where serum CK concentration was assessed with fixed effects for treatment group (categorical variable), visit (ordered categorical variable), and treatment group by visit interaction, and with additional fixed effects for natural log of baseline (continuous variable), screening age covariate (continuous variable), natural log of baseline by visit interaction, and screening age covariate by visit interaction with an unstructured variance-covariance matrix

5. Secondary Outcome: Least Square Mean of Proportion of Skills Gained Based on the Individual Items of the NSAA at Week 52
Description: Proportion of skills gained at Week 52 were expressed as a proportion of the number of skills at Baseline that could be gained (numerator was number of items on NSAA gained at Week 52, with response 1 or 2 and denominator was number of items on NSAA with score 0 at baseline). The NSAA was a 17-item test that graded performance of various functional skills using the following scale: 0 (unable to achieve independently), 1 (modified method but achieves goal independent of physical assistance from another), and 2 ("normal"- no obvious modification of activity). Total score was calculated as the sum of all 17 individual item responses and ranged from 0 (worst) to 34 (fully independent function) with higher scores indicating better function.
Time Frame: Baseline, Week 52
Population: FAS included all eligible participants who were randomly assigned and received a single dose of study drug on Day 1 (Year 1 Day 1). Here, "Overall Number of Participants" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Proportion of skills
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 64 | 26
Proportion of skills | 0.55 [0.41 to 0.68] | 0.42 [0.24 to 0.62]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2; Test type: Superiority; p = 0.2784, Binomial regression; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.64 to 4.62]; The generalized mixed linear model assumed a binomial distribution with logit link & contains fixed effects for treatment group (categorical variable) & screening age (continuous variable)

6. Secondary Outcome: Least Square Mean of Proportion of Skills Either Improved or Maintained Based on the Individual Items of the NSAA at Week 52
Description: Proportion of skills either improved or maintained at Week 52 was expressed as a proportion of the number of items at Baseline that could be improved or maintained (numerator was the number of items on NSAA improved or maintained at Week 52 and denominator is number of items on NSAA which is 17). The NSAA was a 17-item test that graded performance of various functional skills using the following scale: 0 (unable to achieve independently), 1 (modified method but achieves goal independent of physical assistance from another), and 2 ("normal"- no obvious modification of activity). Total score was calculated as the sum of all 17 individual item responses and ranged from 0 (worst) to 34 (fully independent function) with higher scores indicating better function.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Proportion of skills
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 63 | 26
Proportion of skills | 0.88 [0.86 to 0.90] | 0.89 [0.86 to 0.92]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2; Test type: Superiority; p = 0.5437, Binomial Regression; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.63 to 1.28]; The generalized mixed linear model assumed a binomial distribution with a logit link and contained fixed effects for treatment group (categorical variable) and screening age (continuous variable)

7. Secondary Outcome: Change From Baseline in 10 Meter Run/Walk Velocity at Week 52
Description: Velocity was calculated based on the time it took to complete the 10-meter run/walk test.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Meter per second
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 63 | 26
Meter per second | 0.127 [0.039 to 0.215] | 0.206 [0.070 to 0.342]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2; Test type: Superiority; p = 0.3343, Mixed Models Analysis; Least Square Mean Difference = -0.079, 95% CI 2-sided [-0.242 to 0.083], Standard Error of Mean 0.082; The MMRM model contained fixed effects for treatment group (categorical variable), visit (ordered categorical variable), and treatment group by visit interaction with additional fixed effects for baseline value (continuous variable), screening age (continuous variable), baseline value by visit interaction, and screening age by visit interaction with an unstructured variance-covariance matrix

8. Secondary Outcome: Change From Baseline in Rise From Floor Velocity at Week 52
Description: Velocity was calculated based on the time it took to rise from floor.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Meter per second
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 63 | 26
Meter per second | 0.025 [-0.001 to 0.051] | 0.029 [-0.012 to 0.069]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2; Test type: Superiority; p = 0.8826, Mixed Models Analysis; Least Square Mean Difference = -0.004, 95% CI 2-sided [-0.052 to 0.045], Standard Error of Mean 0.024; [other analysis details as in outcome 7, analysis 1]

9. Secondary Outcome: Change From Baseline in Modified Pediatric Outcome Data Collection Instrument (PODCI)- Transfer and Basic Mobility Core Scale at Week 52
Description: Modified PODCI- transfer and basic mobility core scale (parent of pediatric participant) consisted of 11 items that assessed how caregivers of participants evaluated a participant's ability to walk, stand, and perform activities of daily living. The scale produced an independent, standardized score ranging from 0-100, with lower scores representing lower levels of function.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 62 | 27
Score on a scale | 2.18 [0.39 to 3.96] | 0.16 [-2.53 to 2.86]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2; Test type: Superiority; p = 0.2190, Mixed Models Analysis; Least Square Mean Difference = 2.01, 95% CI 2-sided [-1.22 to 5.24], Standard Error of Mean 1.63; [other analysis details as in outcome 7, analysis 1]

10. Secondary Outcome: Change From Baseline in Modified PODCI- Sports and Physical Functioning Core Scale at Week 52
Description: Modified PODCI- sports and physical functioning core scale (parent of pediatric participant) consisted of 21 items that assessed how caregivers of participants evaluated a participant's ability to perform recreational activities. The scale produced an independent, standardized score ranging from 0-100, with lower scores representing lower levels of function.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 62 | 27
Score on a scale | 2.95 [-0.30 to 6.19] | 1.84 [-3.07 to 6.74]
Statistical Analysis 1: Comparison: Cohort 1 vs Cohort 2; Test type: Superiority; p = 0.7096, Mixed Models Analysis; Least Square Mean Difference = 1.11, 95% CI [-4.79 to 7.00], Standard Error of Mean 2.96; [other analysis details as in outcome 7, analysis 1]

ADVERSE EVENTS:
Time Frame: From Year 1 Day 1 up to Week 52
Description: Safety analysis set through Week 52 included all eligible participants who were randomly assigned and received a single dose of study drug on Day 1 (Year 1 Day 1). Same event may appear as both SAE and non-SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/35
Serious Adverse Events (participants affected / at risk) | 25/79 | 5/35
Other Adverse Events (participants affected / at risk) | 77/79 | 20/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=79) | Cohort 2 (N=35)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 3 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 4 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1
Pyrexia (General disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 2 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Troponin I increased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=79) | Cohort 2 (N=35)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 | 0
Abdominal pain (Gastrointestinal disorders) | 17 | 3
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1
Constipation (Gastrointestinal disorders) | 7 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 4
Nausea (Gastrointestinal disorders) | 23 | 3
Vomiting (Gastrointestinal disorders) | 59 | 4
Chest pain (General disorders) | 1 | 2
Fatigue (General disorders) | 7 | 2
Influenza like illness (General disorders) | 0 | 2
Pyrexia (General disorders) | 48 | 3
Ear infection (Infections and infestations) | 4 | 2
Gastroenteritis (Infections and infestations) | 7 | 2
Nasopharyngitis (Infections and infestations) | 19 | 6
Otitis media (Infections and infestations) | 0 | 3
Rhinitis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 7 | 3
Fall (Injury, poisoning and procedural complications) | 4 | 4
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 6 | 0
Glutamate dehydrogenase increased (Investigations) | 19 | 0
Platelet count decreased (Investigations) | 9 | 0
SARS-CoV-2 test positive (Investigations) | 9 | 2
Troponin I increased (Investigations) | 5 | 1
Decreased appetite (Metabolism and nutrition disorders) | 25 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 2
Dizziness (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 13 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 1
Hypertension (Vascular disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-12-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT04281485/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT04281485/SAP_001.pdf